CLINICAL TRIAL: NCT00169156
Title: Study of the Efficacy and the Safety of First Line Treatment With CHOP Plus Rituximab (R-CHOP) in Patients Aged 60 to 80 Years With Previously Untreated T-cell Angioimmunoblastic Lymphoma (AIL).
Brief Title: A Phase II Study of Rituximab Combined With CHOP in T-cell Angio-immunoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAIL; 2005-002602-37 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Untreated T-cell Angioimmunoblastic Lymphoma
Keywords: T-cell angioimmunoblastic lymphoma; Rituximab
MeSH Terms: interventions — Rituximab; Prednisone; Doxorubicin; Cyclophosphamide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab + CHOP (Experimental): Rituximab + CHOP regimen Prednisone - Doxorubicine - Cyclophosphamide - Vincristine
  Interventions: Drug: Rituximab; Drug: Prednisone; Drug: Doxorubicine; Drug: Cyclophosphamide; Drug: Vincristine

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 D1
Drug: Prednisone — 40 mg/m2 D1 to D5
Drug: Doxorubicine — 50 mg/m2 D1
Drug: Cyclophosphamide — 750 mg/m2 D1
Drug: Vincristine — 1,4 mg/m2 D1

SUMMARY:
To evaluate the efficacy and the safety of a front-line treatment combining CHOP regimen and rituximab in patients aged 60 to 80 years with previously untreated AIL.

DETAILED DESCRIPTION:
This is a multicentric, open-label, non-randomized clinical study, evaluating the efficacy and the safety of a front-line treatment combining CHOP regimen and rituximab in patients aged 60 to 80 years with previously untreated AIL.

It is anticipated that 25 subjects will be enrolled over 2 years (from 2005 / 2007).Analysis performed every 5 patients (based on triangular test).

The duration of the treatment period is approximately 25 weeks and patients are followed until Death.

The total Duration of the study is expected to be 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven T-cell angioimmunoblastic lymphoma (AIL) on lymph node biopsy.
* Aged from 60 to 80 years.
* Patient not previously treated (except corticosteroids providing they have been initiated less than 10 days before inclusion).
* ECOG performance status 0 to 2.
* With a minimum of life expectancy > 3 months.
* Negative HIV, HBV and HCV serological tests < 4 weeks (except after vaccination).
* Having previously signed a written informed consent.

Exclusion Criteria:

* Any other histological type of T-cell lymphoma.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug included in the R-CHOP regimen.
* Concurrent severe disease (according to the investigator's decision).
* Active bacterial, viral or fungal infection.
* Poor renal function (serum creatinine level > 150 µmol/L) or impaired liver function tests (total bilirubin level > 30 µmol/L, transaminases > 2.5 upper normal limits) unless they are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils < 1.5 x 109/L or platelets < 100 x 109/L, unless related to bone marrow infiltration.
* Any history of cancer during the last 5 years, with the exception of non basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Patient under tutelage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 8 months (4 cycles of treatment + 4 cycles of consolidation)
  [Complete response (CR), Complete response unconfirmed (CRu)] after the end of treatment.

SECONDARY OUTCOMES:
Event-free survival (EFS) relapse for complete responders, disease progression, early discontinuation of treatment for toxicity or modification of treatment. | 2 years
  Events being death from any cause
Overall survival (OS) | 2 years
Time to progression (TTF) | 2 years
Disease-free survival (DFS). | 2 years
number of SAE | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Haioun, MD, Study Chair — Hôpital Henri Mondor, Créteil, France; Bertrand Joly, MD, Principal Investigator — C.H. Sud Francilien, Corbeil-Essonnes, France
Locations (4):
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attygalle A, Al-Jehani R, Diss TC, Munson P, Liu H, Du MQ, Isaacson PG, Dogan A. Neoplastic T cells in angioimmunoblastic T-cell lymphoma express CD10. Blood. 2002 Jan 15;99(2):627-33. doi: 10.1182/blood.v99.2.627. PMID 11781247
- [Background] Lome-Maldonado C, Canioni D, Hermine O, Delabesse E, Damotte D, Raffoux E, Gaulard P, Macintyre E, Brousse N; French Groupe d'Etude des Lymphomes de l'Adulte (GELA). Angio-immunoblastic T cell lymphoma (AILD-TL) rich in large B cells and associated with Epstein-Barr virus infection. A different subtype of AILD-TL? Leukemia. 2002 Oct;16(10):2134-41. doi: 10.1038/sj.leu.2402642. PMID 12357368
- [Background] Zettl A, Lee SS, Rudiger T, Starostik P, Marino M, Kirchner T, Ott M, Muller-Hermelink HK, Ott G. Epstein-Barr virus-associated B-cell lymphoproliferative disorders in angloimmunoblastic T-cell lymphoma and peripheral T-cell lymphoma, unspecified. Am J Clin Pathol. 2002 Mar;117(3):368-79. doi: 10.1309/6UTX-GVC0-12ND-JJEU. PMID 11888076
- [Background] Gisselbrecht C, Gaulard P, Lepage E, Coiffier B, Briere J, Haioun C, Cazals-Hatem D, Bosly A, Xerri L, Tilly H, Berger F, Bouhabdallah R, Diebold J. Prognostic significance of T-cell phenotype in aggressive non-Hodgkin's lymphomas. Groupe d'Etudes des Lymphomes de l'Adulte (GELA). Blood. 1998 Jul 1;92(1):76-82. PMID 9639502
- See also: Official site of the Groupe d'Etude des Lymphomes de l'Adulte (In french) — http://www.gela.org